CLINICAL TRIAL: NCT05311007
Title: Intrahospital Transport in Patients With High-flow Nasal Oxygenation: Prospective Observational Study.
Acronym: HospiFlow
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2022-01
Record Dates: First submitted 2022-03-23; First posted 2022-04-05 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Critical Illness
Keywords: High-flow nasal oxygenation; intra-hospital transport; critical ill patients; intensive care units
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of the incidence and nature of adverse events — Evaluation of the incidence and nature of adverse events during intra-hospital transport of patients undergoing high-flow nasal oxygen therapy provided by intensive care units

SUMMARY:
High-flow nasal oxygen therapy is commonly used in intensive care unit (ICU). Intra-hospital transfer of critical patients is frequent: 1) to perform diagnostic 2) between emergency room or medical wards and ICU. During theses transfers, oxygenation should be continued.

There is high-flow nasal oxygen therapy for transport using an external battery. This mode of operation in transport mode allows about 30-45 min of autonomy.

Intra-hospital transport under high-flow nasal oxygen therapy has been previously described on children.

The objective of this study is to evaluate the occurrence of complications during intra-hospital transports under high-flow nasal oxygen of critical patients.

DETAILED DESCRIPTION:
High-flow nasal oxygen therapy is commonly used in intensive care unit (ICU). Intra-hospital transfer of critical patients is frequent: 1) to perform diagnostic 2) between emergency room or medical wards and ICU. During theses transfers, oxygenation should be continued.

There is high-flow nasal oxygen therapy for transport using an external battery. This mode of operation in transport mode allows about 30-45 min of autonomy.

Intra-hospital transport under high-flow nasal oxygen therapy has been previously described on children.

The objective of this study is to evaluate the occurrence of complications during intra-hospital transports under high-flow nasal oxygen of critical patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with high-flow nasal oxygen therapy before the intra-hospital transport prior to transport
* Requiring an intra-hospital transport (e.g., CT scan, OR, etc.) or inter-departmental transport supervised by the ICU team

Nb: Once the patient is included in the study, any intra-hospital transport under high-flow nasal oxygen therapy will be analyzed until discharge from the intensive care unit and at until D28.

Exclusion Criteria:

* Under 18 years old
* Patient being under guardianship, tutorship or curatorship
* Pregnancy or breastfeeding
* Lack of social security number
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients requiring intra-hospital transfer on high-flow nasal oxygen therapy will be eligible to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2022-05-28 (Actual); Primary Completion 2024-05-04 (Actual); Study Completion 2024-05-04 (Actual)

PRIMARY OUTCOMES:
Incidence of severe adverse events during intra-hospital transport | Up to 28 days
  To evaluate the incidence of severe adverse events during intra-hospital transport of patients treated with high-flow nasal oxygen surpervised by an ICU staff.
  Severe adverse event is defined by the occurrence of intubation during transport or severe hypoxemia defined as pulse oxygen saturation (SpO2 < 80%) or cardiorespiratory arrest.

SECONDARY OUTCOMES:
Incidence of minor adverse events during intra-hospital transport | Up to 28 days
  To evaluate the incidence of minor adverse events during intra-hospital transport of patients treated with high-flow nasal oxygen surpervised by an ICU staff.
  Minor adverse event is defined by the occurrence of the need to increase the FiO2 or a pull-out of nasal cannulas or the use of an alternative mode of oxygenation (standard oxygen or noninvasive ventilation) or a failure of high-flow nasal oxygenation system (ie battery failure)

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Anh NAY, Dr, Principal Investigator — CHU d'Orléans
Locations (4):
- France (4):
  - Hospital Center of DAX, Dax
  - CH de Martigues, Martigues
  - CHU Orléans, Orléans
  - CH Bretagne Atlantique vannes-Auray, Vannes

REFERENCES:
- [Derived] Nay MA, Bisson A, Auvet A, Delbove A, Berrouba A, Kamel T, Desgrouas M, Boulain T. Intra-hospital transport of adult critically ill patients treated with high flow nasal cannula oxygen: a prospective observational multicenter study. Ann Intensive Care. 2025 Jul 8;15(1):93. doi: 10.1186/s13613-025-01502-7. PMID 40629187